CLINICAL TRIAL: NCT06174896
Title: Comparison of the Airway Sealing Pressures for Three Different Placement Techniques When Using Lma Proseal in Children
Brief Title: LMA Placement Techniques and Airway in Children and Oropharyngeal Leak Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Yasemin Burcu Ustun, Prof.Dr, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: LMAPR1955
Record Dates: First submitted 2023-10-14; First posted 2023-12-18 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Anesthesia; Airway
Keywords: supraglottic airway device; pediatric population
MeSH Terms: interventions — Drug Implants

STUDY DESIGN:
Intervention Model Description: A block randomization list will be created by a doctor who does not participate in patient follow-up using a web-based program, 'Research Randomizer (Urbaniak and Plous 2013)'.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sealed opaque envelopes containing study participation numbers will be used to assign each patient. A researcher not involved in patient follow-up will use the web-based "Research Randomizer" (Urbaniak and Plous 2013) tool to give each participation number to a random group with a 1:1:1 ratio.
  A nurse not an active investigator in the study will have each participant choose an envelope containing the study participation number. They will inform the anesthetist who will administer the methods which group the patient is in immediately before administration. Researchers, patients, surgeons, and nurses will not be aware of the randomization of groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): Placement with standard technique
  Interventions: Procedure: Group 1
- Group 2 (Active Comparator): Placement with direct laryngoscopy
  Interventions: Procedure: Group 2
- Group 3 (Active Comparator): Placement with the aid of video laryngoscopy
  Interventions: Procedure: Group 3

INTERVENTIONS:
Procedure: Group 1 — The LMA Proseal will be inserted directly by hand, without the use of any laryngoscope, as recommended in the instruction manual. The cuff will be gently guided along the hard palate where it is pushed into the hypopharynx and increased resistance is felt, and the cuff will be placed towards the hypopharynx.
  Other Names: Standard technique
  Arms: Group 1
Procedure: Group 2 — Appropriately sized laryngoscope blade will be used and after the location of the epiglottis is determined, the tongue and epiglottis will be lifted forward. Then, LMA Proseal will be placed at the point where resistance is felt at a level where the proximal edge of the mask can be seen.
  Other Names: Placement with direct laryngoscopy
  Arms: Group 2
Procedure: Group 3 — After the video laryngoscope is placed with an appropriately sized blade, the location of the epiglottis and vocal cords will be determined and the LMA Proseal will be placed at the point where slight resistance is encountered after the epiglottis is lifted. proximal aspect of LMA
  Other Names: Placement with the aid of video laryngoscopy
  Arms: Group 3

SUMMARY:
Our study aimed to compare the manual placement, direct laryngoscopy and video laryngoscopy assisted placement techniques of LMA Proseal, a new generation laryngeal mask (LMA), and to find an effective placement technique that does not allow airway leakage in one go.

DETAILED DESCRIPTION:
LMA is an airway device frequently used in pediatric anesthesia. It is preferred for short interventions because it is less invasive compared to intubation. However, problems such as not being fully seated, slipping, and leakage can be encountered during placement. Multiple attempts after unsuccessful placement may cause undesirable results such as edema and sore throat. The aim in this study is to reveal the most accurate placement technique and to transfer this method to clinical applications.

Our research is a prospective, randomized controlled method study.

Patients will be divided into 3 groups.

Group 1:(Standard technique)

Group 2:(Placement with direct laryngoscopy)

Group 3:(Placement with the aid of video laryngoscopy)

After LMA Proseal placement, airway sealing pressures will be measured with appropriate technique. Airway tightness pressure measurement will be made with the technique accepted in the literature through the sensors in the anesthesia machine.

ELIGIBILITY:
Inclusion Criteria:

* 1-10 years old
* Between 5-40 kg
* ASA (American Society of Anesthesiologists) physical score I/II
* Cases undergoing elective surgery lasting less than 90 minutes

Exclusion Criteria:

* Patients who are expected to have a difficult airway
* Those with potential regurgitation risk (severe GER, presence of hiatal hernia)
* Those who will undergo head and neck surgery, laparoscopic surgery
* Those who will undergo surgery in the prone position
* Emergency surgical interventions
* Those who need muscle relaxants
* Presence of intraoral abscess, pharyngeal pathology
* Those who have had an upper or lower respiratory tract infection in the last 4 weeks
* History of allergy to the drugs to be used
* Failure of patients and their relatives to give consent

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure | within 2-3 minutes after laryngeal mask insertion before start of surgery
  Oropharyngeal leak pressure (OLP) will be measured by closing the adjustable pressure limiting valve on the anesthesia machine. The fresh gas flow was adjusted to 3 L/min. When the APL (Adjustable pressure limiting) valve was closed and manually ventilated. The leak sound that occurs during ventilation will be auscultated. The first peak airway pressure at which the leak occurs will be recorded as the oropharyngeal leak pressure.
  After successful insertion, lma proseal location will be evaluated with fiberoptic imaging.

SECONDARY OUTCOMES:
Blood pressure | Preoperatively, one minute after the induction, fifth minute and before removed laryngeal mask.
  Measure blood pressure in millimeter of mercury by non-invasive blood pressure.
İnsertion time | intraoperative period
  LMA insertion time (time from LMA handling to first wave formation in capnography)
Number of placement attempts | intraoperative period
  The number of attempts for optimal placement will be recorded
Need for optimization maneuvers | intraoperative period
  It will be recorded whether additional maneuvering is performed for optimal placement. LMA rotation, jaw thrust, head extension, and flexion will be use as optimization maneuvers.
Complications | intraoperative and postoperative day 1.
  İnvestigate the existence of complications that may be encountered in the routine after LMA placement and removal.
Heart rate | Preoperatively, one minute after the induction, fifth minute and before removed laryngeal mask.
  Measure heart rate in beats per minute by electrocardiography monitor.
Peripheral oxygen saturation | Preoperatively, one minute after the induction, fifth minute and before removed laryngeal mask.
  Measure peripheral oxygen saturation per minute by pulse oximeter.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Burcu Üstün, Prof. Dr, Study Director — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayis University, Samsun, Turkey (Türkiye)

REFERENCES:
- [Background] Oba S, Turk HS, Isil CT, Erdogan H, Sayin P, Dokucu AI. Comparison of the Supreme and ProSeal laryngeal mask airways in infants: a prospective randomised clinical study. BMC Anesthesiol. 2017 Sep 5;17(1):125. doi: 10.1186/s12871-017-0418-z. PMID 28870163
- [Background] Shyam T, Selvaraj V. Airway management using LMA-evaluation of three insertional techniques-a prospective randomised study. J Anaesthesiol Clin Pharmacol. 2021 Jan-Mar;37(1):108-113. doi: 10.4103/joacp.JOACP_60_19. Epub 2021 Apr 10. PMID 34103833
- [Background] Kim GW, Kim JY, Kim SJ, Moon YR, Park EJ, Park SY. Conditions for laryngeal mask airway placement in terms of oropharyngeal leak pressure: a comparison between blind insertion and laryngoscope-guided insertion. BMC Anesthesiol. 2019 Jan 5;19(1):4. doi: 10.1186/s12871-018-0674-6. PMID 30611202